CLINICAL TRIAL: NCT01843192
Title: A Prospective, Multi-Center Evaluation of a Powered Surgical Stapler in Video-Assisted Thoracoscopic Lung Resection Procedures
Brief Title: Powered Echelon Device in VATS Surgery
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC-12-001
Record Dates: First submitted 2013-04-19; First posted 2013-04-30 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VATS for suspected or confirmed NSCLC: Single arm study
  Interventions: Device: Endocutter

INTERVENTIONS:
Device: Endocutter

SUMMARY:
This study aims to collect real world outcomes of Video-Assisted Thoracoscopic Surgery (VATS) for lung cancer (lobectomy, wedge resection) using ECHELON FLEX™ Powered ENDOPATH® Staplers 45 mm and/or 60 mm (study devices).

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed NSCLC (up to and including Stage II)
* Scheduled for lung resection surgery (lobectomy or wedge resection) involving only one lobe of the lung
* Performance status 0-1 (Eastern Cooperative Oncology Group classification)
* ASA score < 3
* No prior history of VATS or open lung surgery
* Willing to give consent and comply with study-related evaluation and treatment schedule

Exclusion Criteria:

* Active bacterial infection or fungal infection;
* Systemic administration (intravenous or oral) of steroids (within 30 days prior to study procedure)
* Chemotherapy or radiation therapy for lung cancer may not be performed for 30 days prior to the procedure
* Scheduled concurrent surgical procedure other than wedge resection or lobectomy (central venous access - e.g. port placement, mediastinoscopy with lymph node sampling, and VATS lymphadenectomy are allowed)
* Pregnancy
* Physical or psychological condition which would impair study participation;
* The patient is judged unsuitable for study participation by the Investigator for any other reason; or
* Unable or unwilling to attend follow-up visits and examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with suspected or confirmed NSCLC, scheduled for VATS lobectomy or wedge resection in accordance with their institution's SOC
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Dignity Health, St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals undergoing VATS lobectomy for suspected or confirmed Non-small Cell Lung Cancer, or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of Care, and who meet study entry criteria, were enrolled in this study.
Pre-assignment Details: There was no assignment to treatment group given that this is a single arm study wherein the same device was used on all subjects. Results are presented for the overall cohort as well as by the individual procedure performed - lobectomy, wedge resection, or wedge resection with lobectomy.
Groups:
- Wedge Resection: Subjects undergoing VATS wedge resection
- Lobectomy: Subjects undergoing VATS lobectomy
- Wedge Resection With Lobectomy: Subjects undergoing VATS wedge resection that also required lobectomy
Period: Overall Study
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Started | 26 | 34 | 11
Completed | 24 | 28 | 9
Not Completed | 2 | 6 | 2
Not completed — Intra-operative exclusions per protocol | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Population: All subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure
Groups:
- Total: Total of all reporting groups
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy | Total
Number analyzed (Participants) | 24 | 28 | 9 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.02) | 68.1 (7.26) | 68.7 (5.72) | 66.3 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 20 | 5 | 37
  Male | 12 | 8 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 28 | 9 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 23 | 27 | 9 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 9 | 61

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Postoperative Air Leaks
Description: Air leak was to be quantitatively assessed starting on the evening after surgery and then twice daily (during morning and evening rounds) as described by Certfolio et al. 2001. Patients were instructed to perform standardized repeated forced expiratory maneuvers (coughing and blowing). Leaks were scored using the air-leak meter that comes as part of a pleura vac system from 1 to 7, with 7 being the highest (most chambers).
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
percentage of participants | 45.8 [25.6 to 67.2] | 67.9 [47.6 to 84.1] | 88.9 [51.8 to 99.7]

2. Primary Outcome: Occurrence of Prolonged Air Leaks
Description: Prolonged air leaks defined as longer than 5 days in continuous duration. Air leak was to be quantitatively assessed starting on the evening after surgery and then twice daily (during morning and evening rounds) as described by Certfolio et al. 2001. Patients were instructed to perform standardized repeated forced expiratory maneuvers (coughing and blowing). Leaks were scored using the air-leak meter that comes as part of a pleura vac system from 1 to 7, with 7 being the highest (most chambers).
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
percentage of participants | 4.2 [0.1 to 21.1] | 7.1 [0.9 to 23.5] | 22.2 [2.8 to 60]

3. Secondary Outcome: Length of Stay (LOS)
Description: Determined as the length of time in days from hospital admission to initial hospital discharge
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
days | 3.7 (1.63) | 4.9 (1.70) | 4.8 (1.48)

4. Secondary Outcome: Volume of Estimated Intra-operative Blood Loss
Time Frame: Blood loss intra-op and up to 5 days post-op
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
milliliters | 31.5 (56.48) | 83.2 (62.42) | 86.1 (80.15)

5. Secondary Outcome: Time to Chest Tube Removal
Description: Defined as the number of days from date of surgery to removal of the last chest tube inserted during the surgical procedure.
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
days | 3.7 (1.63) | 4.9 (1.7) | 4.8 (1.48)

6. Secondary Outcome: Operative Time
Description: Defined as the duration in hours from the first skin incision to the closure of the last incision
Time Frame: Day of surgery
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
hours | 1.7 (0.68) | 2.8 (0.85) | 3.4 (1.43)

7. Secondary Outcome: Occurrence of Intra-operative Leak Test
Description: This outcome was scored as Yes or No based on whether a leak was detected during an intra-operative leak test when it was performed. Not all subjects had an intra-operative leak test performed, as it was not standard of care at all participating institutions, and so results are only presented for those subjects in whom an intra-operative test was performed.
Time Frame: During surgery
Population: All subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure. This analysis was further restricted to those subjects in whom an intra-operative leak test was actually performed, as it was not standard of care at all participating institutions.
Measure: Number; unit: participants
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 2 | 12 | 3
participants | 0 | 0 | 1

8. Secondary Outcome: Number of Subjects With 1 Chest Tube Placed
Description: All subjects had either 1 or 2 chest tubes placed during surgery. Results presented are for the percentage of subjects with 1 chest tube placed.
Time Frame: During surgery
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 24 | 28 | 9
percentage of participants | 88.5 | 100 | 88.9

ADVERSE EVENTS:
Time Frame: Duration of follow-up was scheduled through approximately 4 weeks post surgery
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Serious Adverse Events (participants affected / at risk) | 2/26 | 4/34 | 2/11
Other Adverse Events (participants affected / at risk) | 8/26 | 6/34 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wedge Resection (N=26) | Lobectomy (N=34) | Wedge Resection With Lobectomy (N=11)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wedge Resection (N=26) | Lobectomy (N=34) | Wedge Resection With Lobectomy (N=11)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Vascular injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less